CLINICAL TRIAL: NCT00895895
Title: A 52-Week, Two-Period, Multicenter, Randomized, Double-Blind, Donepezil-Referenced, Placebo-Controlled, Efficacy And Safety Study Of 3 Dosage Levels Of SAM-531 In Outpatients With Mild To Moderate Alzheimer Disease
Brief Title: Study Comparing 3 Dosage Levels Of SAM-531 In Outpatients With Mild To Moderate Alzheimer Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3193A1-2005; B1961007; NCT01312896 (obsolete NCT alias)
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): SAM-531 1.5 mg
  Interventions: Drug: SAM-531 1.5 mg
- 3 (Experimental): SAM-531 3.0 mg
  Interventions: Drug: SAM-531 3.0 mg
- 4 (Experimental): SAM-531 5.0 mg
  Interventions: Drug: SAM-531 5.0 mg
- 5 (Active Comparator): Donepezil
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Placebo — Capsules SAM-531 placebo and 5 mg tablet encapsulated Donepezil placebo capsules, once a day during 24 weeks.
  Arms: 1
Drug: SAM-531 1.5 mg — Capsules SAM-531 1.5 mg, once a day during 52 weeks.
  Arms: 2
Drug: SAM-531 3.0 mg — Capsules SAM-531 3.0 mg, once a day during 52 weeks.
  Arms: 3
Drug: SAM-531 5.0 mg — Capsules SAM-531 5.0 mg, once a day during 24 weeks or 52 weeks.
  Arms: 4
Drug: Donepezil — Encapsulated Donepezil 5 mg tablets, once a day during 52 weeks. After Day 42, the dose can up titrated up to 10 mg of Donepezil.
  Arms: 5

SUMMARY:
The study will evaluate the efficacy and safety of an investigational drug called SAM-531 at three dosage levels. Subjects will receive either one of the 3 dosage levels of SAM-531, donepezil or placebo for the first 24 weeks of the study (period I). Subjects who receive placebo for period I will be assigned to receive the highest dose of SAM-531 SAM-531 for the remaining 28 weeks of the study, while subjects who received one of the three SAM-531 dosage levels or donepezil in period I will continue with the same study drug (period II).

DETAILED DESCRIPTION:
The study was stopped (date of termination was 13April2011) due to a 6 month interim analysis: all of the 3 SAM-531 dosage levels were declared futile. There were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer Disease according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Diseases and Related Disorders Association (NINCDS-ADRDA) criteria.
* Mini-Mental State Examination (MMSE) score of 12 to 24 at screening
* Rosen Modified Hachinski Ischemic score < or equal to 4 at screening.

Exclusion Criteria:

* Relevant neurologic disease other than Alzheimer Disease that may affect cognition or ability to complete the study.
* Current major depressive disorder or other current major psychiatric disorder.
* History of clinically evident stroke or clinically important carotid or vertebrobasilar stenosis or plaque.
* Use of prescription or nonprescription medications for cognitive enhancement (including memantine, ginkgo biloba, huperzine A, and cholinesterase inhibitors) within 3 months before the baseline visit.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (78):
- United States (31):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Oxnard, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Atlantis, Florida
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Elk Grove Village, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Cedarhurst, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Bennington, Vermont
  - Pfizer Investigational Site, Middleton, Wisconsin
- Argentina (3):
  - Pfizer Investigational Site, C.a.b.a., Buenos Aires
  - Pfizer Investigational Site, Caba, Buenos Aires
  - Pfizer Investigational Site, Ciudad de Buenos Aires
- Chile (2):
  - Pfizer Investigational Site, Santiago, Chile
  - Pfizer Investigational Site, Viña del Mar, Chile
- Colombia (5):
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Pereira, Risaralda Department
  - Pfizer Investigational Site, Bucamaranga, Santander Department
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
  - Pfizer Investigational Site, Valle Del Cauca
- Hong Kong (2):
  - Pfizer Investigational Site, Shatin, N.T., Hong Kong SAR, China
  - Pfizer Investigational Site, Hong Kong
- Japan (10):
  - Pfizer Investigational Site, Hachiōji, Tokyo
  - Pfizer Investigational Site, Chiba
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Hiroshima
  - Pfizer Investigational Site, Kanagawa
  - Pfizer Investigational Site, Kumamoto
  - Pfizer Investigational Site, Kyoto
  - Pfizer Investigational Site, Nagano
  - Pfizer Investigational Site, Nagasaki
  - Pfizer Investigational Site, Shizuoka
- Mexico (2):
  - Pfizer Investigational Site, Saltillo, Coahuila
  - Pfizer Investigational Site, Aguascalientes
- New Zealand (2):
  - Pfizer Investigational Site, Auckland
  - Pfizer Investigational Site, Hamilton
- Poland (4):
  - Pfizer Investigational Site, Krakow, Poland
  - Pfizer Investigational Site, Poznan, Poland
  - Pfizer Investigational Site, Wroclaw, Poland
  - Pfizer Investigational Site, Krakow
- Romania (3):
  - Pfizer Investigational Site, Craiova, Dolj
  - Pfizer Investigational Site, Timișoara, Timiș County
  - Pfizer Investigational Site, Bucharest
- Russia (7):
  - Pfizer Investigational Site, Nikolskoe Village, Gatchina District, Leningrad Region
  - Pfizer Investigational Site, Kazan'
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Novosibirsk
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk
  - Pfizer Investigational Site, Yaroslavl
- South Africa (5):
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Bellville, Western Cape
  - Pfizer Investigational Site, Cape Town
- South Korea (2):
  - Pfizer Investigational Site, Seongnam-si, Gyeonggi-do
  - Pfizer Investigational Site, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3193A1-2005&StudyName=Study%20Comparing%203%20Dosage%20Levels%20Of%20SAM-531%20In%20Outpatients%20With%20Mild%20To%20Moderate%20Alzheimer%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then SAM-531: Matching SAM-531 placebo capsule administered orally once daily (QD, morning) and matching encapsulated Donepezil placebo tablet QD (evening) for up to 24 weeks (Period 1). Then from Week 25 up to Week 52 (Period 2) participants received SAM-531 5.0 milligram (mg) capsule administered once daily (QD, morning) and matching encapsulated Donepezil placebo tablet administered QD (evening). From Week 7 until Week 52 (end of study), the evening dose in both period 1 and 2 could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 (1.5 mg): SAM-531 1.5 mg capsule administered orally QD (morning) for up to 52 weeks. Matching encapsulated Donepezil placebo tablet administered QD (evening) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 (3.0 mg): SAM-531 3.0 mg capsule administered orally QD (morning) for up to 52 weeks. Matching encapsulated Donepezil placebo tablet administered orally QD (evening) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 (5.0 mg): SAM-531 5.0 mg capsule administered orally QD (morning) for up to 52 weeks. Matching encapsulated Donepezil placebo tablet administered orally QD (evening) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- Donepezil: Matching SAM-531 placebo capsule administered orally (QD, morning) for up to 52 weeks. Encapsulated Donepezil 5 mg tablet administered orally (QD, evening) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
Period: Period 1
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Started | 107 | 105 | 104 | 104 | 106
Randomized But Not Treated | 1 | 3 | 1 | 1 | 2
Completed | 86 | 84 | 84 | 91 | 86
Not Completed | 21 | 21 | 20 | 13 | 20
Not completed — Adverse Event | 7 | 6 | 4 | 6 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — discontinued by sponsor | 2 | 1 | 2 | 1 | 1
Not completed — failed to return | 0 | 0 | 1 | 0 | 1
Not completed — investigator request | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 3 | 2 | 3
Not completed — Other | 1 | 2 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 8 | 2 | 4
Not completed — unsatisfactory response-efficacy | 2 | 0 | 0 | 0 | 0
Not completed — randomized and not treated | 1 | 3 | 1 | 1 | 2
Period: After Period 1, Prior to Period 2
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Started | 86 | 84 | 84 | 91 | 86
Completed | 86 | 84 | 82 | 91 | 84
Not Completed | 0 | 0 | 2 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Started | 86 | 84 | 82 | 91 | 84
Completed | 30 | 31 | 33 | 37 | 35
Not Completed | 56 | 53 | 49 | 54 | 49
Not completed — Adverse Event | 3 | 3 | 5 | 2 | 5
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — discontinued by sponsor | 44 | 44 | 38 | 46 | 37
Not completed — failed to return | 2 | 0 | 0 | 0 | 0
Not completed — investigator request | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 1 | 0
Not completed — Other | 1 | 1 | 3 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 3 | 5
Not completed — unsatisfactory response-efficacy | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil | Total
Number analyzed (Participants) | 106 | 102 | 103 | 103 | 104 | 518
Age, Customized [Number; unit: participants]
  50 to 65 years | 22 | 17 | 19 | 18 | 20 | 96
  66 to 80 years | 59 | 60 | 54 | 66 | 66 | 305
  greater than 80 years | 25 | 25 | 30 | 19 | 18 | 117
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 70 | 71 | 73 | 70 | 356
  Male | 34 | 32 | 32 | 30 | 34 | 162

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale-Cognition (ADAS-Cog) Total Score at Week 24
Description: 14-item scale to assess severity of cognitive impairment in Alzheimer's Disease. Items: word recall, naming objects and fingers, following commands, constructional praxis, ideational praxis, orientation, word recognition, recall of test instructions, spoken language ability, word-finding difficulty, comprehension of spoken language, concentration/distractibility, number cancellation and executive maze. Rating scale ranged from 0 (not present) to 5 (severe). Total score was sum of individual scores (items 1-11) and ranged from 0 to 70 with higher scores indicating greater cognitive impairment.
Time Frame: Baseline, Week 24
Population: Intent to treat (ITT) population: randomized participants who took at least one dose of study medication, had a baseline evaluation and had at least one on-treatment post-baseline evaluation for the ADAS-Cog; Number of Participants Analyzed (N): number of evaluable participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 99 | 98 | 100 | 101 | 103
units on a scale
  Baseline | 23.6 (10.3) | 24.1 (11.7) | 23.6 (10.6) | 22.6 (9.8) | 23.4 (10.0)
  Week 24 | 23.8 (12.0) | 24.2 (13.1) | 23.5 (12.0) | 21.9 (10.6) | 22.4 (10.9)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.424, Mixed Models Analysis; Mixed Model with repeated measures: change=Mini Mental State Examination (MMSE) Japan baseline baseline times(*)visit visit treatment treatment*visit; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.0 to 2.3]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.849, Mixed Models Analysis; Mixed Model with repeated measures: change equals (=) MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.8 to 1.5]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.520, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-2.2 to 1.1]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.258, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.6 to 0.7]

2. Secondary Outcome: Change From Baseline in Disability Assessment for Dementia (DAD) Total Score at Week 24
Description: Caregiver interview-based instrument assessing 10 areas of activities of daily living (ADL) to measure participant's actual performance over the previous 2 weeks. Items included hygiene, dressing, continence, eating, meal preparation, telephoning, outings, finance/correspondence, medications and leisure/housework. Responses scored as 1 (yes) or 0 (no), response of "Not Applicable" was not scored. Total DAD score was sum of scores for 40 items, expressed as a percentage of the number of items answered yes or no. Total score ranged from 0 to 100, higher scores represented less disability in ADL.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: percentage of yes answers
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 97 | 97 | 98 | 100 | 102
percentage of yes answers
  Baseline | 77.4 (21.8) | 73.1 (20.9) | 72.9 (22.5) | 75.5 (21.0) | 73.2 (22.9)
  Week 24 | 76.7 (24.2) | 71.4 (25.0) | 73.0 (24.4) | 76.8 (23.1) | 75.6 (24.5)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.367, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-5.2 to 1.9]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.910, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-3.3 to 3.7]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.160, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-1.0 to 6.0]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.060, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-0.1 to 6.9]

3. Secondary Outcome: Change From Baseline in Neuropsychiatry Inventory (NPI) at Week 24
Description: Caregiver interview-based rating scale assessed 10 behavioral, 2 neurovegetative disturbances occurring in dementia: delusions, hallucination, agitation/aggression, depression, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability, aberrant motor behavior, appetite/eating disorders and sleep/nightime behavior disorders. Each symptom score derived by symptom frequency (1 [occasionally] to 4 [very frequently] * symptom severity (1 [mild] to 3 [severe]) and ranged 0-12. Total score = sum of symptom scores; range 0-144, higher score indicating greater behavioral disturbances
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 96 | 96 | 98 | 99 | 102
unit on a scale
  Baseline | 10.6 (13.9) | 14.6 (16.6) | 14.8 (18.1) | 13.4 (13.4) | 12.1 (14.8)
  Week 24 | 10.7 (14.4) | 11.9 (14.6) | 9.7 (11.3) | 10.4 (11.4) | 9.3 (12.9)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.931, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.8 to 3.1]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.054, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-5.8 to 0.1]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.246, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-4.6 to 1.2]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.426, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-4.1 to 1.7]

4. Secondary Outcome: Number of Participants With Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) Scores at Week 24
Description: Caregiver and participant interview-based tool to rate the overall impression of participant's clinical change of the disease over time. Areas covered in the interview include: relevant history, observation/evaluation, mental/cognitive state, behavior and functioning. Change categorized into 1 of 7 categories: marked improvement, moderate improvement, minimal improvement, no change, minimal worsening, moderate worsening, marked worsening.
Time Frame: Baseline, Week 24
Population: ITT; N=number of evaluable participants
Measure: Number; unit: participants
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 86 | 85 | 84 | 92 | 87
participants
  marked improvement | 0 | 1 | 1 | 1 | 1
  moderate improvement | 1 | 2 | 5 | 3 | 4
  minimal improvement | 20 | 23 | 19 | 17 | 23
  no change | 32 | 36 | 33 | 45 | 30
  minimal worsening | 30 | 17 | 19 | 22 | 25
  moderate worsening | 2 | 5 | 6 | 4 | 3
  marked worsening | 1 | 1 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg) vs SAM-531 (3.0 mg) vs SAM-531 (5.0 mg) vs Donepezil; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Test type: Superiority or Other; p = 0.682, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Test type: Superiority or Other; p = 0.532, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo, Then SAM-531 vs Donepezil; Test type: Superiority or Other; p = 0.751, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in Cambridge Neuropsychological Test Automated Battery (CANTAB) Paired Associate Learning (PAL)Total Errors (N, Shapes, Adjusted) at Week 24
Description: CANTAB PAL-assessed visual memory/new learning using one or more patterns randomly displayed in boxes on a screen. Participants were to touch the box where patterns first appeared. Stage 1 (practice) and difficulty increased Stage 2 (2 patterns) to Stage 6 (6 patterns). When all locations correctly identified moved to next Stage. Test terminated when a stage could not be completed in 6 attempts. Total Errors=total number of incorrect boxes chosen plus adjustment for estimated possible errors on problems, attempts, and recalls not reached. Total score 0 to 106, lower scores=better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 94 | 93 | 97 | 96 | 98
errors
  Baseline | 68.3 (27.4) | 66.9 (29.6) | 66.5 (28.6) | 67.6 (28.8) | 67.8 (29.3)
  Week 24 | 66.4 (27.4) | 68.1 (29.2) | 67.5 (29.8) | 64.9 (30.8) | 66.7 (28.6)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.553, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-3.9 to 7.3]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.886, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-6.0 to 5.2]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.712, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-6.6 to 4.5]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.785, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-4.8 to 6.4]

6. Secondary Outcome: Change From Baseline in CANTAB PAL - Number of Patterns Reached at Week 24
Description: CANTAB PAL-assessed visual memory/new learning using one or more patterns randomly displayed in boxes on a screen. Participants were to touch the box where patterns first appeared. Stage 1 (practice) and difficulty increased Stage 2 (2 patterns) to Stage 6 (6 patterns). When all locations correctly identified moved to next Stage. Test terminated when a stage could not be completed in 6 attempts. Total score was the number of patterns presented at last stage successfully completed and ranged from 2 to 6, higher scores indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: patterns
Groups:
- SAM-531 (1.5 mg): SAM-531 1.5 mg capsule administered orally QD (morning) for up to 52 weeks. Matching Donepezil placebo tablet administered QD (evening) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 94 | 93 | 97 | 96 | 98
patterns
  Baseline | 4.1 (1.3) | 4.2 (1.3) | 4.2 (1.3) | 4.1 (1.4) | 4.1 (1.3)
  Week 24 | 4.3 (1.3) | 4.1 (1.4) | 4.2 (1.4) | 4.2 (1.5) | 4.2 (1.4)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.251, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.993, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.553, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.611, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2]

7. Secondary Outcome: Change From Baseline in CANTAB PAL - First Trial Memory Score, Patterns at Week 24
Description: CANTAB PAL-assessed visual memory/new learning using one or more patterns randomly displayed in boxes on a screen. Participants were to touch the box where patterns first appeared. Stage 1 (practice) and difficulty increased Stage 2 (2 patterns) to Stage 6 (6 patterns). When all locations correctly identified moved to next Stage. Test terminated when a stage could not be completed in 6 attempts. Total score was the number of correct choices made on the first attempt at each Stage. Total score ranged from 0 to 20, higher scores indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: correct choices
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 94 | 93 | 97 | 96 | 98
correct choices
  Baseline | 4.6 (3.9) | 4.8 (4.5) | 4.7 (4.3) | 4.6 (4.1) | 4.6 (4.4)
  Week 24 | 4.8 (4.0) | 4.4 (4.2) | 4.8 (4.5) | 5.1 (4.5) | 4.5 (4.1)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.340, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.5 to 0.5]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.630, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.8 to 1.2]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.678, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.8 to 1.2]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.518, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.3 to 0.7]

8. Secondary Outcome: Change From Baseline in CANTAB Spatial Working Memory (SWM) - Between Errors (4 Boxes) at Week 24
Description: CANTAB-SWM assessed participant's retention of spatial information, ability to manipulate remembered items and strategize. Participant asked to find tokens in on-screen boxes, move them. Difficulty ranged 4-8 boxes to assess, 2 trials per assessment. Between errors: number of times participant revisited a box where a token previously found. In 4 box assessments the maximum number of errors per trial was 20. Test ended with 20 errors in a trial. Less than 20 errors in both trials the participant went to the next level of difficulty. Scores ranged from 0 to 39. Lower scores: better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 95 | 93 | 97 | 97 | 98
errors
  Baseline | 3.8 (2.0) | 3.6 (2.4) | 3.8 (2.7) | 3.5 (2.1) | 3.9 (2.4)
  Week 24 | 3.7 (2.3) | 3.6 (2.3) | 3.7 (2.5) | 3.1 (2.3) | 3.5 (2.3)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.953, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.956, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.216, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.2]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.665, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.5]

9. Secondary Outcome: Change From Baseline in CANTAB-SWM - Between Errors (6 Boxes) at Week 24
Description: CANTAB-SWM assessed participant's retention of spatial information, ability to manipulate remembered items and strategize. Participant asked to find tokens in on-screen boxes, move them. Difficulty ranged 4-8 boxes to assess, 2 trials per assessment. Between errors: number of times participant revisited a box where a token previously found. In 6 box assessments the maximum number of errors per trial was 30. Test ended with 30 errors in a trial. Less than 30 errors in both trials the participant went to the next level of difficulty. Scores ranged from 0 to 59. Lower scores: better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 95 | 93 | 97 | 97 | 98
errors
  Baseline | 9.2 (3.9) | 9.1 (4.2) | 9.1 (3.9) | 8.6 (4.0) | 10.0 (4.8)
  Week 24 | 8.9 (2.9) | 9.2 (4.9) | 9.0 (4.1) | 9.1 (3.9) | 8.9 (3.7)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.373, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.6 to 1.7]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.781, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.0 to 1.3]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.417, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.7 to 1.6]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.853, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.3 to 1.0]

10. Secondary Outcome: Change From Baseline in CANTAB SWM - Between Errors (8 Boxes) at Week 24
Description: CANTAB-SWM assessed participant's retention of spatial information, ability to manipulate remembered items and strategize. Participant asked to find tokens in on-screen boxes, move them. Difficulty ranged 4-8 boxes to assess, 2 trials per assessment. Between errors: number of times participant revisited a box where a token previously found. In 8 box assessments the maximum number of errors per trial was 40. Test ended with 40 errors in a trial. Less than 40 errors in both trials the participant went to the next level of difficulty. Scores ranged from 0 to 79. Lower scores: better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 95 | 93 | 97 | 97 | 98
errors
  Baseline | 20.7 (5.9) | 20.1 (5.8) | 20.8 (6.1) | 19.3 (6.9) | 20.2 (6.5)
  Week 24 | 21.1 (5.6) | 20.0 (6.4) | 20.8 (5.4) | 19.7 (7.1) | 19.8 (5.8)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.428, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.6 to 1.1]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.763, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.1 to 1.5]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.312, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.7 to 0.9]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.215, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.0 to 0.7]

11. Secondary Outcome: Change From Baseline in CANTAB SWM - Between Errors (N Boxes) at Week 24
Description: CANTAB-SWM assessed participant's retention of spatial information, ability to manipulate remembered items and strategize. Participant was asked to find tokens in on-screen boxes and move them. Difficulty ranged from 4 to 8 box assessments, 2 trials for each assessment. Possible errors for each successful assessment: 4 box 0-38; 6 box 0-58; 8 box 0-78. Between Errors for N Boxes was the cumulative number of errors per each successful trial. Total scores ranged from 0 to 175. Lower scores indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 95 | 93 | 97 | 97 | 98
errors
  Baseline | 33.8 (9.0) | 32.8 (9.4) | 33.7 (10.0) | 31.4 (8.9) | 34.2 (10.4)
  Week 24 | 33.8 (7.8) | 32.8 (10.3) | 33.5 (9.6) | 32.0 (10.2) | 32.2 (9.5)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.956, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.7 to 2.5]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.988, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-2.6 to 2.5]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.890, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.7 to 2.4]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.280, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.0 to 1.2]

12. Secondary Outcome: Change From Baseline in CANTAB SWM Strategy at Week 24
Description: CANTAB-SWM assessed participant's ability to strategize. Participant was asked to find tokens in on-screen boxes and move them. Difficulty ranged from 4 to 8 box assessments, 2 trials per assessment. Strategy score was the number of unique boxes the participant searched in the two 6 and 8 box trials. 6 box trial scores ranged from 1 (1 box searched for all 6 tokens) to 6 (6 boxes searched for 6 tokens). 8 box trial score ranged from 1 (1 box searched) to 8 (8 boxes searched for 8 tokens). Total of the 4 trial scores ranged from 4 to 28. Lower score indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: boxes
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 95 | 93 | 97 | 97 | 98
boxes
  Baseline | 19.7 (3.1) | 19.4 (3.3) | 19.2 (2.8) | 19.1 (3.6) | 19.0 (3.6)
  Week 24 | 20.0 (2.2) | 19.1 (3.3) | 19.4 (2.3) | 19.0 (3.9) | 20.0 (2.0)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.154, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.5 to 0.2]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.740, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.0 to 0.7]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.179, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.4 to 0.3]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.543, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.6 to 1.1]

13. Secondary Outcome: Change From Baseline in CANTAB Pattern Recognition Memory (PRM)-Mean Correct Latency at Week 24
Description: CANTAB-PRM assessed participant's visual pattern recognition memory in a 2-choice forced discrimination paradigm. Participants presented with a series of 12 visual patterns singly. In recognition phase, participants were required to choose between a pattern previously seen and a novel pattern. Patterns in the recognition phase appeared sequentially in reverse order on the screen. Assessment was repeated with 12 new patterns. Latency in correct responses ranged from 0 to infinity millisecond (msec), lower scores indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 95 | 96 | 97 | 98 | 99
msec
  Baseline | 4583.7 (3121.2) | 4121.1 (2358.8) | 4973.4 (2784.3) | 4216.4 (2208.6) | 4303.0 (2705.2)
  Week 24 | 4288.3 (2082.7) | 3979.1 (3002.3) | 3793.5 (1698.0) | 4301.5 (2931.4) | 4387.8 (2703.8)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.861, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -60.4, 95% CI 2-sided [-739.7 to 618.8]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -926.6, 95% CI 2-sided [-1596.9 to -256.3]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.676, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 141.3, 95% CI 2-sided [-522.1 to 804.6]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.505, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 230.6, 95% CI 2-sided [-449.7 to 910.9]

14. Secondary Outcome: Change From Baseline in CANTAB PRM-Percentage Correct at Week 24
Description: CANTAB-PRM assessed participant's visual pattern recognition memory in a 2-choice forced discrimination paradigm. Participants presented with a series of 12 visual patterns singly. In recognition phase, participants were required to choose between a pattern previously seen and a novel pattern. Patterns in the recognition phase appeared sequentially in reverse order on the screen. Assessment was repeated with 12 new patterns. Correct response total expressed as a percentage, ranged from 0 to 100, higher scores indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 95 | 96 | 97 | 98 | 99
percentage of correct answers
  Baseline | 59.3 (18.7) | 62.2 (18.4) | 63.4 (17.1) | 66.7 (17.7) | 63.9 (18.9)
  Week 24 | 59.4 (16.3) | 63.0 (20.2) | 64.4 (18.4) | 65.9 (17.6) | 63.7 (16.9)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.267, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-2.2 to 7.8]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.145, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-1.3 to 8.6]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.139, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-1.2 to 8.6]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.386, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-2.8 to 7.2]

15. Secondary Outcome: Change From Baseline in CANTAB Reaction Time (RTI) Five-Choice Accuracy at Week 24
Description: CANTAB-RTI assessed participant's reaction, movement time and vigilance during a 5-choice reaction time trial and to measure anticipatory/premature and perseverative responses. In the trial, a yellow spot appeared on a computer screen in 1 of 5 locations, the participant responded by letting go of a press pad and touching the screen where the spot appeared. 5-Choice Accuracy was the total number of trials where participant responded correctly. Total ranged from 0 to 30, higher score indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: correct trials
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 89 | 93 | 96 | 96 | 95
correct trials
  Baseline | 27.3 (4.4) | 26.9 (5.8) | 27.0 (5.6) | 28.1 (4.4) | 27.0 (5.4)
  Week 24 | 27.8 (3.2) | 26.7 (5.9) | 28.1 (4.0) | 28.1 (3.4) | 27.9 (4.6)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.032, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.3 to -0.1]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.264, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.5 to 1.7]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.893, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.0 to 1.1]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.525, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.7 to 1.4]

16. Secondary Outcome: Change From Baseline in CANTAB RTI Five-Choice Movement Time at Week 24
Description: CANTAB-RTI assessed participant's reaction, movement time and vigilance during 5-choice reaction time trial and also measured anticipatory/premature responses. In the test, a yellow spot appeared on a computer screen in 1 of 5 locations, the participant responded by letting go of a press pad and touching the screen where the spot appeared. 5-Choice Movement Time was the time from release of press pad to screen touch where the spot had been in trials the participant responded correctly. Possible score ranged from 100 to 5100 msec, lower score indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 88 | 93 | 96 | 96 | 95
msec
  Baseline | 573.5 (218.6) | 583.1 (307.5) | 617.6 (381.9) | 564.4 (310.0) | 583.6 (292.8)
  Week 24 | 539.9 (199.0) | 578.8 (290.9) | 584.7 (284.9) | 546.4 (191.0) | 560.6 (284.6)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 60.9, 95% CI 2-sided [-1.6 to 123.5]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.488, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 21.8, 95% CI 2-sided [-40.0 to 83.5]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.783, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [-52.6 to 69.8]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.578, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 17.6, 95% CI 2-sided [-44.6 to 79.8]

17. Secondary Outcome: Change From Baseline in CANTAB RTI Five-Choice Reaction Time at Week 24
Description: CANTAB-RTI assessed participant's reaction, movement time and vigilance during 5-choice reaction time trial and also measured anticipatory/premature responses. In the test, a yellow spot appeared on a computer screen in 1 of 5 locations, the participant responded by letting go of a press pad and touching the screen where the spot appeared. 5-Choice Reaction Time was the time from appearance of yellow spot on computer screen to time to release press pad in trials the participant responded correctly. Total ranged from 100 to 5100 (maximum allowed) msec, lower score indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 88 | 93 | 96 | 96 | 95
msec
  Baseline | 488.6 (275.8) | 503.7 (215.2) | 488.6 (200.8) | 438.2 (172.1) | 475.7 (205.9)
  Week 24 | 447.3 (139.3) | 483.6 (211.3) | 473.7 (184.4) | 438.5 (170.7) | 443.3 (145.5)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 31.1, 95% CI 2-sided [-13.9 to 76.1]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.352, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 21.0, 95% CI 2-sided [-23.3 to 65.4]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.797, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-38.1 to 49.6]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.633, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-55.6 to 33.9]

18. Secondary Outcome: Change From Baseline in CANTAB RTI Simple Movement Time at Week 24
Description: CANTAB-RTI assessed participant's reaction, movement time and vigilance during simple (1 choice) reaction time trial and also measured anticipatory/premature responses. In the test, 1 yellow spot appeared on a computer screen in 1 location, the participant responded by letting go of a press pad and touching the screen where the spot appeared. Simple Movement Time was the time from release of press pad to touch the screen where the spot had been in trials the participant responded correctly. Total ranged from 100 to 5100 (maximum allowed) msec, lower score indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 89 | 92 | 96 | 96 | 95
msec
  Baseline | 620.4 (299.0) | 631.2 (379.2) | 669.0 (473.8) | 641.2 (443.0) | 624.0 (336.0)
  Week 24 | 585.2 (253.2) | 630.6 (359.5) | 641.8 (366.4) | 604.6 (262.2) | 621.0 (331.8)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 71.2, 95% CI 2-sided [-4.7 to 147.0]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.598, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 20.0, 95% CI 2-sided [-54.6 to 94.7]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.766, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 11.2, 95% CI 2-sided [-62.9 to 85.3]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.378, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 33.8, 95% CI 2-sided [-41.5 to 109.1]

19. Secondary Outcome: Change From Baseline in CANTAB RTI Simple Reaction Time at Week 24
Description: CANTAB-RTI assessed participant's reaction, movement time and vigilance during simple (1 choice) reaction time trial and also measured anticipatory/premature responses. In the test, 1 yellow spot appeared on a computer screen in 1 location, the participant responded by letting go of a press pad and touching the screen where the spot appeared. Simple Reaction Time was the time from appearance of yellow spot on computer screen to time to release press pad in trials the participant responded correctly. Total ranged from 100 to 5100 (maximum allowed) msec, lower score indicated better performance.
Time Frame: Baseline, Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 89 | 92 | 96 | 96 | 95
msec
  Baseline | 471.8 (219.7) | 510.9 (295.1) | 487.1 (255.1) | 442.8 (247.3) | 501.3 (302.9)
  Week 24 | 449.2 (195.8) | 479.7 (327.7) | 460.4 (213.5) | 445.3 (206.0) | 445.5 (203.6)
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.481, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 22.5, 95% CI 2-sided [-40.2 to 85.2]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.894, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-57.5 to 65.9]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.991, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-61.5 to 60.8]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Analysis of adjusted difference in change from baseline; Test type: Superiority or Other; p = 0.422, Mixed Models Analysis; Mixed Model with repeated measures: change = MMSE Japan baseline baseline * visit visit treatment treatment * visit; Mean Difference (Final Values) = -25.5, 95% CI 2-sided [-87.9 to 36.9]

20. Secondary Outcome: Percentage of Participants Who Were Responders at Week 24
Description: Responder defined as a participant who demonstrated an improvement of at least 3 points from baseline in the ADAS-Cog total score and no worsening in the DAD total score and in ADCS-CGIC. Participants were considered a responder at Week 24 if all 3 criteria were met.
Time Frame: Week 24
Population: ITT; N=number of participants with evaluable data
Measure: Number; unit: percentage of participants
Arm/Group | Placebo, Then SAM-531 | SAM-531 (1.5 mg) | SAM-531 (3.0 mg) | SAM-531 (5.0 mg) | Donepezil
Number analyzed (Participants) | 87 | 85 | 86 | 92 | 87
percentage of participants | 9.2 | 7.1 | 10.5 | 15.2 | 20.7
Statistical Analysis 1: Comparison: Placebo, Then SAM-531 vs SAM-531 (1.5 mg); Test type: Superiority or Other; p = 0.581, Regression, Logistic; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.24 to 2.22]
Statistical Analysis 2: Comparison: Placebo, Then SAM-531 vs SAM-531 (3.0 mg); Test type: Superiority or Other; p = 0.770, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.42 to 3.19]
Statistical Analysis 3: Comparison: Placebo, Then SAM-531 vs SAM-531 (5.0 mg); Test type: Superiority or Other; p = 0.216, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.71 to 4.55]
Statistical Analysis 4: Comparison: Placebo, Then SAM-531 vs Donepezil; Test type: Superiority or Other; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.06 to 6.42]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Placebo/5.0 mg Period 1: Matching SAM-531 placebo capsule administered QD (morning dose) and one encapsulated Donepezil placebo tablet administered QD (evening dose) for up to 24 weeks (Period 1). From Week 7 the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 1.5 mg Period 1: SAM-531 1.5 mg capsule administered QD (morning dose) through 24 weeks. Matching encapsulated Donepezil placebo tablet administered QD (evening dose) through 24 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 3.0 mg Period 1: SAM-531 3.0 mg capsule administered QD (morning dose) through 24 weeks. Matching encapsulated Donepezil placebo tablet administered QD (evening dose) through 24 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 5.0 mg Period 1: SAM-531 5.0 mg capsule administered QD (morning dose) through 24 weeks. Matching encapsulated Donepezil placebo tablet administered QD (evening dose) through 24 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- Donepezil Period 1: Matching SAM-531 placebo capsule administered QD (morning dose) and 1 encapsulated Donepezil 5 mg tablet administered orally QD (evening dose) through 24 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion and according to tolerance.
- SAM-531 5.0 mg Crossover Period 2: Participants who received Placebo in Period 1, beginning in Week 25 and up to Week 52 (Period 2) received SAM-531 5.0 mg capsule administered QD (morning dose) and matching encapsulated Donepezil placebo tablet administered QD (evening dose). The evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 1.5 mg Period 2: SAM-531 1.5 mg capsule administered QD (morning dose) Week 25 up to 52 weeks. Matching encapsulated Donepezil placebo tablet administered QD (evening dose) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 3.0 mg Period 2: SAM-531 3.0 mg capsule administered QD (morning dose) Week 25 up to 52 weeks. Matching encapsulated Donepezil placebo tablet administered QD (evening dose) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- SAM-531 5.0 mg Period 2: SAM-531 5.0 mg capsule administered QD (morning dose) Week 25 up to 52 weeks. Matching encapsulated Donepezil placebo tablet administered QD (evening dose) for up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion.
- Donepezil Period 2: Matching SAM-531 placebo capsule administered QD (morning dose) for up to 52 weeks. One encapsulated Donepezil 5 mg tablet administered orally QD (evening dose) from Week 25 up to 52 weeks. From Week 7 until Week 52 (end of study), the evening dose could have been increased to 2 tablets and adjusted back to 1 tablet at the investigator's discretion and according to tolerance.
Arm/Group | Placebo/5.0 mg Period 1 | SAM-531 1.5 mg Period 1 | SAM-531 3.0 mg Period 1 | SAM-531 5.0 mg Period 1 | Donepezil Period 1 | SAM-531 5.0 mg Crossover Period 2 | SAM-531 1.5 mg Period 2 | SAM-531 3.0 mg Period 2 | SAM-531 5.0 mg Period 2 | Donepezil Period 2
Serious Adverse Events (participants affected / at risk) | 7/106 | 7/102 | 8/103 | 4/103 | 4/104 | 8/106 | 2/102 | 7/103 | 3/103 | 7/104
Other Adverse Events (participants affected / at risk) | 30/106 | 23/102 | 32/103 | 37/103 | 24/104 | 13/106 | 13/102 | 22/103 | 22/103 | 19/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/5.0 mg Period 1 (N=106) | SAM-531 1.5 mg Period 1 (N=102) | SAM-531 3.0 mg Period 1 (N=103) | SAM-531 5.0 mg Period 1 (N=103) | Donepezil Period 1 (N=104) | SAM-531 5.0 mg Crossover Period 2 (N=106) | SAM-531 1.5 mg Period 2 (N=102) | SAM-531 3.0 mg Period 2 (N=103) | SAM-531 5.0 mg Period 2 (N=103) | Donepezil Period 2 (N=104)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/5.0 mg Period 1 (N=106) | SAM-531 1.5 mg Period 1 (N=102) | SAM-531 3.0 mg Period 1 (N=103) | SAM-531 5.0 mg Period 1 (N=103) | Donepezil Period 1 (N=104) | SAM-531 5.0 mg Crossover Period 2 (N=106) | SAM-531 1.5 mg Period 2 (N=102) | SAM-531 3.0 mg Period 2 (N=103) | SAM-531 5.0 mg Period 2 (N=103) | Donepezil Period 2 (N=104)
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 4 | 9 | 7 | 0 | 2 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 5 | 1 | 6 | 2 | 3 | 1 | 0 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5 | 2 | 6 | 5 | 3 | 3 | 2 | 8 | 4
Urinary tract infection (Infections and infestations) | 7 | 4 | 11 | 2 | 3 | 5 | 3 | 8 | 5 | 2
Dizziness (Nervous system disorders) | 0 | 5 | 7 | 3 | 2 | 0 | 1 | 3 | 1 | 2
Headache (Nervous system disorders) | 6 | 6 | 8 | 11 | 4 | 2 | 2 | 7 | 4 | 5
Insomnia (Psychiatric disorders) | 3 | 1 | 2 | 8 | 1 | 1 | 3 | 1 | 4 | 4
Hypertension (Vascular disorders) | 6 | 2 | 3 | 4 | 4 | 4 | 2 | 5 | 1 | 3

LIMITATIONS AND CAVEATS:
Study terminated early due to futility. Period 2 events include those that started in Period 2 or started in Period 1 and continued in to Period 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.